CLINICAL TRIAL: NCT06166134
Title: Radiological Evaluation of Sarcopenia in Patient Received Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Maher, Resident doctor, Assiut University
Other Study IDs: Us and CT in sarcopenia
Record Dates: First submitted 2023-12-02; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiological evaluation of sarcopenia in patients receiving chemotherapy

DETAILED DESCRIPTION:
Evaluation of muscle mass by using sonoelastography and computed tomography

ELIGIBILITY:
Inclusion Criteria:

* all cancer patients receiving chemotherapy referred to radiodiagnosis department for routine examination Patients must be between 18 and

Exclusion Criteria:

* Previous or current history of any musculoskeletal or neurological disorder including strokes.
* Systemic atrophy affecting CNS ( Huntington disease ,hereditary ataxia ,spinal muscular disorder and related syndromes ,post polio syndrome )
* Central nervous system demyelinating disease ( Multiple sclerosis , acute disseminated demyelinated syndromes..
* Corticosteroids undertaken currently or for the past 3 years with doses >5mg/day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Comparison of muscle mass before and after chemotherapy by use of sonoelastography and computed tomography and comparison with normal volunteer
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Radiological evaluation of sarcopenia in patients receiving chemotherapy | April 2025
  Using sonoelastography and computed tomography in evaluation of muscle mass in patients received chemotherapy by measurement of muscle thickness ,echogencity ,cross sectional area ,fasicle length,pennation angle, strain ratio,shear wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Refaat, Assisstant professor, Study Director — Assiut university -south egypt cancer institute; Omar Mostafa, Assisstant professor, Study Director — Assiut university -south egypt cancer institute

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36227071/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35054402/